CLINICAL TRIAL: NCT06263686
Title: Prospective, Randomized, Double-blind Parallel Group Nutritional Study to Evaluate the Effects of Routine Intake of Fresh vs- Pasteurized Yoghurt on the Immune System in Healthy Adults
Brief Title: Evaluation of the Effects of Routine Intake of Fresh vs- Pasteurized Yoghurt on the Immune System in Healthy Adults
Acronym: YASI-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Danone Institute International (Other); University of Seville (Other)
Responsible Party: Principal Investigator, Alfredo Corell, Proffesor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DAN056
Record Dates: First submitted 2024-01-17; First posted 2024-02-16 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Immune System; Innate Inflammatory Response
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pasteurised yoghurt (Experimental)
  Interventions: Other: Pasteurised yoghurt
- Fresh natural yoghurt (Experimental)
  Interventions: Other: Fresh yoghurt
- Sterilised yoghurt (Experimental)
  Interventions: Other: Sterilised yoghurt

INTERVENTIONS:
Other: Pasteurised yoghurt — Pasteurised (heat treated) natural yoghurt containing <15 CFU/g of Lactobacillus delbrueckii bulgacirus and <15 CFU/g of Streptococcus thermophilus.
  Arms: Pasteurised yoghurt
Other: Fresh yoghurt — containing ≥ 108 CFU/g of Lactobacillus delbrueckii bulgacirus and ≥ 108 CFU/g of Streptococcus thermophilus
  Arms: Fresh natural yoghurt
Other: Sterilised yoghurt — Not containing viable bacteria
  Arms: Sterilised yoghurt

SUMMARY:
In this study, the purpose was to describe and compare the modulator effects on the immune system of the routine ingestion of fresh vs. pasteurized yoghurt. A unicentral, prospective, randomized, double-blind, parallel group nutritional study for 8 weeks was carried out comparing the ingestion of 125 g (three times a day) of the products in healthy adults. A complete battery of in vitro tests on the activity of immune system, processes and phenomena was performed.

ELIGIBILITY:
Inclusion criteria

* Age between 20 and 70 years, both included.
* Healthy or mildly ill subjects (without any current chronic pharmacotherapy).
* Body mass index between 18.5 and 29.9 kg/m2, both included.
* Subjects who usually follow a balanced diet that are not engaged in any therapeutic lifestyle change involving stringent dietary interventions such as weight-reducing diets.
* Written informed consent to participate

Exclusion criteria

* Patients could not meet any the following criteria at the screening visit to be included in the study.
* Subjects with diseases or disorders affecting the function of the immune system, such as auto-immune diseases, allergies, atopic conditions, hypersensitivity to any kind of stimulus, or immunosupression for any reason; even if they are not currently taken any pharmacotherapy.
* Subjects with relevant functional or structural disorder affecting the gastrointestinal tract, such as malformations, angiodysplasias, active peptic ulcers or chronic inflammatory disease of the intestine; even if they are not in any specific pharmacotherapy at the time of recruitment; or who have underwent surgical procedures with permanent sequels (for example, gastroenterostomy).
* Subjects with any infectious disease requiring antibiotherapy at the time of recruitment.
* Subjects following any treatment modifying the immune response, such as immunosuppressants, corticosteroids, etc.
* Subjects with celiac disease.
* Subjects with chronic background weakening conditions, such as diabetes or neoplasms.
* Subjects with history of renal lithiasis.
* Subjects with deficient nutritional or hydrational status.
* Subjects with relevant deviations in routine haematology or biochemistry parameters.
* Subjects with current and documented alcohol abuse.
* Subjects in whom the investigator expected insufficient collaboration or difficulties to follow the study procedures.
* Subjects who regularly took any of the forbidden products specified in the appropriate section.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
T-cells | Up to 6 weeks
  T-cells measured as percentage of CD3 positive cells among the blood lymphocytes (defined by gating as CD45 bright and low cellular complexity or side scatter)
IFN-gamma induction | Up to 6 weeks
  T-lymphocyte function: stimulation with PHA and measurement of Intracellular synthesis of IFN-γ in terms of percentage of IFN producing cells among the CD3 CD4 double positive (T helper cells)
IgG | Up to 6 weeks
  serum IgG concentration measured in mg/dl

REFERENCES:
- [Result] Rivero-Pino F, Casquete M, Castro MJ, Redondo Del Rio P, Gutierrez E, Mayo-Iscar A, Nocito M, Corell A. Prospective, Randomized, Double-Blind Parallel Group Nutritional Study to Evaluate the Effects of Routine Intake of Fresh vs. Pasteurized Yogurt on the Immune System in Healthy Adults. Nutrients. 2024 Jun 20;16(12):1969. doi: 10.3390/nu16121969. PMID 38931322